CLINICAL TRIAL: NCT06824766
Title: Investigation of the Relationship Between Autonomic Nervous System Activity and Biomechanical Characteristics of Chewing Muscles in Bruxers
Brief Title: Chewing Muscles in Bruxers
Status: Recruiting | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Hazel Çelik Güzel, Assist. Prof. Dr, Bandırma Onyedi Eylül University
Other Study IDs: 2024-248
Record Dates: First submitted 2025-02-05; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Bruxism
Keywords: Autonomic nervous system; bruxism; masseter
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Bruxers: Individuals with bruxism
  Interventions: Other: Visual Analogue Scale; Other: Autonomic nervous system activity assessment; Other: Masticatory muscles assessment
- Control group: Healthy volunteers
  Interventions: Other: Visual Analogue Scale; Other: Autonomic nervous system activity assessment; Other: Masticatory muscles assessment

INTERVENTIONS:
Other: Visual Analogue Scale — The pain intensity of the participants will be assessed using the Visual Analogue Scale, which is a simple, reliable and short-term method commonly used to measure pain intensity in the clinic. The participant is told that the most severe pain he/she experiences is 10 and if there is no pain, the pain intensity is 0. The participant will be asked to tick a number between 0 and 10 corresponding to the intensity of pain felt in the masticatory muscles at rest and during chewing.
Other: Autonomic nervous system activity assessment — All participants included in the study will undergo a 5-minute test with the Polar H10 chest strap device for autonomic nervous system activity assessment (heart rate variability assessment). The data obtained after the measurement will be analysed with Kubios software. Stress index (cardiovascular system stress), PNS index (parasympathetic nervous system dominance), SNS index (sympathetic nervous system dominance), LF power (sympathetic activity), HF power (parasympathetic activity) and LF/HF ratio (sympathetic/parasympathetic balance) parameters will be used in the evaluation of HRV in Kubios programme.
Other: Masticatory muscles assessment — The Myoton PRO device will be used to objectively assess the biomechanical properties of the participants' masticatory muscles such as tone, stiffness and elasticity. The masseter and temporalis muscles will be evaluated bilaterally in the sitting position. Three measurements will be recorded at one second intervals and the average value will be used for analysis.

SUMMARY:
The aim of this study was to determine the relationship between autonomic nervous system activity and tonus, stiffness and elasticity of temporalis and masseter muscles in individuals with bruxism and to compare them with healthy controls.

DETAILED DESCRIPTION:
Individuals diagnosed with bruxism and healthy individuals as a control group will be included in the study. Firstly, the purpose of the research and evaluation methods will be explained to the participants. Individuals who volunteer to participate in the study and meet the inclusion criteria will be included. Approval will be obtained from the individuals to be evaluated with the 'Informed Voluntary Consent Form'. Individuals will then fill in the Descriptive Data Form. The intensity of pain in the masticatory muscles of all participants at rest and during chewing will be measured by Visual Analogue Scale, Autonomic Nervous System activity (heart rate variables) will be measured by Polar H10 chest strap, and the tonus, stiffness and elasticity of the temporalis and masseter muscles will be measured by Myoton device. The evaluations are planned to take an average of 20 minutes for each participant. The evaluations of the participants will be made only once and will not be evaluated again.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with bruxism between the ages of 18-65,
* A history of bruxism for at least 6 months,
* Individuals with masseter muscle pain ≥4 at rest and during mastication
* Control group: Healthy individuals aged 18-65 years

Exclusion Criteria:

* Masseter botox application in the last 6 months,
* With regular use of analgesics and anti-inflammatories affecting the OSS,
* Smokes 20 or more cigarettes daily,
* With regular alcohol use of 1-2 glasses per day,
* Daily coffee consumption of 6 cups or more,
* Cardiovascular, respiratory and central nervous system diseases,
* Presence of infection or tumoural structures within intraoral structures,
* Multiple ear piercings,
* With TMJ disc displacement and joint degeneration,
* Cervical or TMJ fracture, systemic disease, musculoskeletal problem with evidence of specific pathological condition,
* Any surgical operation related to cervical or TMJ problem,
* Less than 6 months of cervical or TMJ-related physiotherapy and rehabilitation services,
* The one with facial paralysis,
* Diagnosed psychiatric illness
* Participants who have communication difficulties in speaking and understanding Turkish or who are unable to understand the exercises

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bruxers
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | March 1, 2025- June 1, 2025
  The pain intensity of the participants will be assessed using the Visual Analogue Scale, which is a simple, reliable and short-term method commonly used to measure pain intensity in the clinic. The participant is told that the most severe pain he/she experiences is 10 and if there is no pain, the pain intensity is 0. The participant will be asked to tick a number between 0 and 10 corresponding to the intensity of pain felt in the masticatory muscles at rest and during chewing.
Autonomic nervous system activity assessment | March 1, 2025- June 1, 2025
  All participants included in the study will undergo a 5-minute test with the Polar H10 chest strap device for autonomic nervous system activity assessment. The data obtained after the measurement will be analysed with Kubios software.
Masticatory muscles biomechanical properties assessment | March 1, 2025- June 1, 2025
  The Myoton PRO device will be used to objectively assess the biomechanical properties of the participants' masticatory muscles. The masticatory muscles will be evaluated bilaterally in the sitting position. Three measurements will be recorded at one second intervals and the average value will be used for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylül University, Balıkesir, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided